CLINICAL TRIAL: NCT04382300
Title: Safety and Efficacy of Pyrotinib Combined With Thalidomide in Advanced Non-Small-Cell Lung Cancer With HER2 Exon 20 Insertions: A Prospective, Single-arm, Open-label Phase II Study
Brief Title: Pyrotinib Plus Thalidomide in Advanced NSCLC Patients Harboring HER2 Exon 20 Insertions
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Lu Shun, Director of the Oncology department, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-NSCLC-II-005
Record Dates: First submitted 2020-04-30; First posted 2020-05-11 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Non-small-cell Lung Cancer
Keywords: Pyrotinib; HER2; Non-small-cell Lung Cancer; Phase II; Thalidomide
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Thalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): pyrotinib 400mg p.o. qd, combined with thalidomide 200mg p.o. qd
  Interventions: Drug: pyrotinib combined with thalidomide

INTERVENTIONS:
Drug: pyrotinib combined with thalidomide — Single Group Assignment

SUMMARY:
Various driver gene mutations have been identified in lung cancer. Among them, human epidermal growth factor 2 (HER2) was identified in approximately 2% of non-small-cell lung cancers. Pyrotinib is an oral tyrosine kinase inhibitor targeting both HER-1 and HER-2 receptors. This is a prospective, single-arm, open-label phase II study, designed to evaluate the efficacy and safety of pyrotinib combined with thalidomide in advanced non-small-cell lung cancer patients with HER2 exon 20 insertions.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years.
* ECOG performance status 0-1.
* Life expectancy ≥12 weeks.
* At least one measurable lesion according to RECIST 1.1.
* Histologically or cytologically confirmed advanced (IIIB or IV) non-small-cell lung cancer according to the 7th edition of TNM classification and staging system for lung cancer published by IASLC.
* HER2 exon 20 insertions confirmed by next generation sequencing or polymerase chain reaction (if blood samples are used, the mutation abundance should be ≥10%).
* Disease progression during or after platinum-based chemotherapy, or refusing chemotherapy (patients are allowed to have prior therapy with PD-1/PD-L1 inhibitors and/or antiangiogenic agents).
* No more than two prior chemotherapy regimens (a. replacing platinum drug due to toxicity is considered as a new regimen; b. adjuvant chemotherapy is not considered as a prior regimen if disease recurrence occurred at more than 6 months after the last dose).
* No radiotherapy within 3 months, or prior radiotherapy with radiation area <25% of bone marrow area at least 4 weeks before enrollment.
* Required laboratory values including following parameters:

ANC: ≥ 1.5 × 10^9/L, Platelet count: ≥ 90 × 10^9/L, Hemoglobin: ≥ 90 g/L, INR: ≤1.5, APTT: ≤1.5 × ULN, Total bilirubin: ≤ 1.5 × ULN, ALT and AST: ≤ 2 × ULN for liver metastases, BUN and creatine: ≤ 1.5 × ULN, creatine clearance rate: ≥ 50 mL/min, LVEF: ≥ 50%, QTcF: < 470 ms for female, < 450 ms for male.

* Willingness to use highly effective contraception from the start of the study to 90 days after the last dose of study drug.
* Written informed consent.

Exclusion Criteria:

* Prior HER2-targeting therapies.
* Other gene alterations with available targeted drugs, such as EGFR mutations, T790M resistance mutations, ALK fusions, ROS1 fusions, RET rearrangements, BRAF V600E mutations, NTRK fusions, and MET exon 14 skipping.
* Factors influencing the oral administration of drugs, such as inability to swallow, chronic diarrhea, intestinal obstruction, or other gastrointestinal diseases or abnormalities.
* With third space effusion that can not be controlled by drainage or other methods.
* Radiotherapy, chemotherapy, surgery, or other targeted therapy for non-small-cell lung adenocarcinoma within 4 weeks.
* Active brain metastases, meningeal metastases, spinal compression, or CT or MRI revealing brain or leptomeningeal diseases at screening (patients with symptomatically stable brain metastases can be enrolled if no cerebral hemorrhage is found by brain MRI, CT or venography).
* Uncontrolled hypokalemia or hypomagnesemia.
* Allergy history to the components of study drug.
* History of immunodeficiency disease (including positive test of human immunodeficiency virus, active hepatitis B/C, or other acquired or congenital immunodeficiency disease) or organ transplantation.
* History of cardiac diseases, including angina, arrhythmia requiring drug therapy or of clinical significance, myocardial infarction, heart failure, and other cardiac diseases unsuitable for this trial as judged by the investigator.
* Patients with thrombotic disease or previous history of thrombosis.
* Other malignancies within 5 years, except for cured cervical cancer in situ, skin basal cell cancer, and skin squamous cell cancer.
* History of neurological or mental disorders, such as epilepsy and dementia.
* Respiratory syndrome (dyspnea ≥grade 2 using NCI CTCAE 5.0).
* Coagulation disorders (INR >1.5, prothrombin time >ULN + 4 s, or APTT >1.5×ULN), with bleeding tendency or receiving thrombolytic or anticoagulant therapy.
* Renal dysfunction (urine protein ≥++, or 24-hour proteinuria ≥1.0 g).
* Participating in other clinical trials within 4 weeks.
* Pregnant or lactating woman.
* Concomitant diseases seriously affecting the patient safety or the completion of study as judged by the investigator, such as uncontrolled severe hypertension, severe diabetes mellitus, and active infection.
* Any other condition unsuitable for the study as judged by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 24 months
  The proportion of patients with complete response or partial response.

SECONDARY OUTCOMES:
Progression-free Survival | 24 months
  Time from the initiation of treatment to disease progression or death, whichever came first.
Overall Survival | 24 months
  Time from the initiation of treatment to death.
Disease Control Rate | 24 months
  The proportion of patients with complete response, partial response or stable disease.
Incidence of Adverse Events | 24 months
  Adverse events was graded according to NCI CTCAE 5.0.
Changes in Scores of European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) | 24 months
  QLQ-C30 scores were standardized to a scale ranging from 0-100 by linear transformation. For global health status/quality of life and functional subscales, higher scores indicate a higher (better) level of function, whereas for the symptom subscales, higher scores indicate a higher (worse) severity of symptoms.
Changes in Scores of EORTC Quality of Life Questionnaire-Lung Cancer Module 13 (QLQ-LC13) | 24 months
  QLQ-LC13 scores were standardized to a scale ranging from 0-100 by linear transformation. For global health status/quality of life and functional subscales, higher scores indicate a higher (better) level of function, whereas for the symptom subscales, higher scores indicate a higher (worse) severity of symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology, Shanghai Lung Cancer Center, Shanghai Chest Hospital, Shanghai Jiao Tong University, Shanghai, China

REFERENCES:
- [Derived] Ai X, Song Z, Jian H, Zhou Z, Chen Z, Yu Y, Li Z, Lu S. Pyrotinib combined with thalidomide in advanced non-small-cell lung cancer patients harboring HER2 exon 20 insertions (PRIDE): protocol of an open-label, single-arm phase II trial. BMC Cancer. 2021 Sep 16;21(1):1033. doi: 10.1186/s12885-021-08759-8. PMID 34530760